CLINICAL TRIAL: NCT05463926
Title: Effectiveness of 'Parentbot - a Digital Healthcare Assistant (PDA)', a Mobile Application-based Intervention, in Improving Parental Psychosocial Outcomes During the Perinatal Period: a Randomized Controlled Trial and Process Evaluation
Brief Title: Effect of 'Parentbot - a Digital Healthcare Assistant (PDA)' in Improving Parenting Outcomes During the Perinatal Period
Acronym: PDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Shefaly Shorey, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NHG DSRB 2021/00227
Record Dates: First submitted 2022-07-14; First posted 2022-07-19 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Perinatal Depression; Parents; Self Efficacy; Anxiety; Stress; Parenting Satisfaction
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Two-group parallel-armed randomized controlled trial (RCT) with a pretest and repeated posttest experimental design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard hospital care with follow-up + PDA mobile application (Experimental): Receive standard hospital care and follow-up, and access to the Parentbot - a Digital healthcare Assistant (PDA) mobile application from pregnancy until one-month postpartum
  Interventions: Behavioral: PDA mobile application
- Standard hospital care with follow-up (No Intervention): Receive standard hospital care with follow-up

INTERVENTIONS:
Behavioral: PDA mobile application — Parentbot - a Digital healthcare Assistant (PDA):
  A mobile application-based psychosocial parenting intervention with integrated chatbot features. It consists of multimedia educational materials (text files, audio files and videos), discussion forums, guided mindfulness-based meditation videos, guided reflection and gratitude journals and a chatbot.
  Arms: Standard hospital care with follow-up + PDA mobile application

SUMMARY:
The Parentbot - a Digital healthcare Assistant (PDA) is a mobile application-based psychosocial parenting intervention with integrated chatbot features, intended for couples to use during the perinatal period. It provides parents with multimedia educational materials (text files, audio files and videos), discussion forum, guided mindfulness-based meditation videos, guided reflection and gratitude journals and a chatbot to answer their queries related to perinatal care in real-time.

This study aims to:

1. Develop a theory-based perinatal intervention with integrated chatbot features for both first-time and experienced parents
2. Examine the effectiveness of the PDA intervention in improving parenting self-efficacy (primary outcome), stress, depression, anxiety, social support, parent-child bonding and parenting satisfaction (secondary outcomes) among parents during the perinatal period
3. Examine the perceptions of parents from both the intervention and control group after the intervention
4. Collate suggestions for further improvement from the participants and members of the research team

The hypotheses of this study are:

The PDA intervention group will have significantly higher scores for parenting self-efficacy, social support, parent-child bonding and parenting satisfaction, as well as lower scores for stress, depression and anxiety compared to the control group receiving standard care after the intervention at one-month postpartum (post-test 1) and three-months postpartum (post-test 2).

ELIGIBILITY:
Inclusion Criteria:

Heterosexual married couples who are first-time parents or experienced parents are included if they:

* Are at least 21 years old
* Are fluent in English
* Own a smartphone with internet access
* Intend to stay in Singapore until three months postpartum
* Are having a low-risk singleton or multiple pregnancy at > 24 gestational weeks (age of viability).

Exclusion Criteria:

Couples will be excluded if either parent has:

* Any self-reported psychiatric disorders, visual, auditory, cognitive impairment and/or any major medical condition that can affect their abilities to participate in the trial
* High-risk pregnancy including placenta previa major, pre-eclampsia, intrauterine growth restriction etc
* Suffer from a miscarriage or made the decision to abort their child
* Give birth to still-birth newborn
* Give birth to a newborn with congenital anomalies or medical complications (require intensive care, severe jaundice, Down's syndrome)

Single parents will also be excluded. If either the mother or father declines to participate in the study while their partner agrees, the couple will not be allowed to participate in the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Parenting self-efficacy | 1 month postpartum
  10-item Parenting Efficacy Scale (PES): Score ranges from 10-40, with higher scores indicating a higher level of perceived parenting self-efficacy
Parenting self-efficacy | 3 months postpartum
  10-item Parenting Efficacy Scale (PES): Score ranges from 10-40, with higher scores indicating a higher level of perceived parenting self-efficacy

SECONDARY OUTCOMES:
Stress | 1 month postpartum
  10-item Perceived Stress Scale (PSS): Score ranges from 0-40, with higher scores indicating higher stress levels
Stress | 3 months postpartum
  10-item Perceived Stress Scale (PSS): Score ranges from 0-40, with higher scores indicating higher stress levels
Depression | 1 month postpartum
  10-item Edinburgh Postnatal Depression Scale (EPDS) Scale: Score ranges from 0-30, with higher scores indicating more severe depressive symptoms
Depression | 3 months postpartum
  10-item Edinburgh Postnatal Depression Scale (EPDS) Scale: Score ranges from 0-30, with higher scores indicating more severe depressive symptoms
Anxiety | 1 month postpartum
  40-item State-Trait Anxiety Inventory (STAI): Score ranges from 40-160, with higher scores indicating more severe anxiety symptoms
Anxiety | 3 months postpartum
  40-item State-Trait Anxiety Inventory (STAI): Score ranges from 40-160, with higher scores indicating more severe anxiety symptoms
Social support | 1 month postpartum
  4-item Perceived Social Support for Parenting scale (PSSP): Score ranges from 0-16, with higher scores indicating higher level of perceived social support
Social support | 3 months postpartum
  4-item Perceived Social Support for Parenting scale (PSSP): Score ranges from 0-16, with higher scores indicating higher level of perceived social support
Parent-child bonding | 1 month postpartum
  8-item Parent-Infant Bonding Questionnaire (PIBQ): Score ranges from 0-24, with higher scores indicating poorer parent-child bonding
Parent-child bonding | 3 months postpartum
  8-item Parent-Infant Bonding Questionnaire (PIBQ): Score ranges from 0-24, with higher scores indicating poorer parent-child bonding
Parenting satisfaction | 1 month postpartum
  11-item evaluation subscale of the What Being the Parent of a Baby is Like scale (WBPL): Score ranges from 0-90, with higher scores indicating greater parenting satisfaction
Parenting satisfaction | 3 months postpartum
  11-item evaluation subscale of the What Being the Parent of a Baby is Like scale (WBPL): Score ranges from 0-90, with higher scores indicating greater parenting satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Shefaly Shorey, PhD, Principal Investigator — National University of Singapore
Locations (1):
- Alice Lee Centre for Nursing Studies, National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chua JYX, Choolani M, Chee CYI, Yi H, Chan YH, Lalor JG, Chong YS, Shorey S. The effectiveness of Parentbot - a digital healthcare assistant - on parenting outcomes: A randomized controlled trial. Int J Nurs Stud. 2024 Dec;160:104906. doi: 10.1016/j.ijnurstu.2024.104906. Epub 2024 Sep 13. PMID 39305680